CLINICAL TRIAL: NCT00757419
Title: A Phase 1 Single Centre Single-blind Randomised Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral AZD3355 After Administration of Single Ascending Doses and Multiple Repeated Doses in Healthy Male Volunteers
Brief Title: AZD3355 Dose-escalation Study in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Debra G. Silberg, MD, PhD, Medical Science Director, AZD3355, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D9120C00030; EudraCTnr: 2008-003578-16
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Reflux Disease
Keywords: Safety; tolerability; healthy subjects
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — lesogaberan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD3355
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3355 — capsules, oral, single or twice daily dose
  Other Names: Lesogaberan
  Arms: 1
Drug: Placebo — To match dosing of AZD3355
  Arms: 2

SUMMARY:
The aim is to establish the maximal tolerated dose of AZD3355 for the selection of doses in the up-coming studies. This will be done by comparing single and repeated doses of AZD3355 to placebo ("inactive substance"). Safety and tolerability variables will be closely monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects without concurrent diseases who do not require any medical treatments
* Provision of signed informed consent.

Exclusion Criteria:

* History of somatic disease/condition, which may interfere with the objectives for the study, as judged by the investigator.
* Clinically significant illness or clinically relevant trauma within the 2 weeks prior to the administration of the investigational product, as judged by the investigator.
* History of clinically significant orthostatic reaction or syncope
* Clinically important abnormalities related to the heart function

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety variables (Adverse event reporting, ECG, blood pressure, pulse rate, urine weight and osmolality, body temperature, blood and urine laboratory values) | During the study

SECONDARY OUTCOMES:
Pharmacokinetic variables | Several occasions during the study days

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Hartford, Principal Investigator — CPU Avd 102, Gröna Stråket 12, Sahlgrenska Universitetssjukhuset, 413 45 Göteborg; Eva Ersdal, Study Director — AstraZeneca R&D, Mölndal, Sweden
Locations (1):
- Research Site, Gothenburg, Sweden